CLINICAL TRIAL: NCT03662347
Title: Patient Acceptable Symptomatic State and Minimal Clinically Important Difference of the Fatigue in Multiple Sclerosis (SeDiF_SEP)
Acronym: SeDiF_SEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00403-52; APJC2016/SeDIF_SEP-EPSTEIN/AS (Other: sponsor code)
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fatigue is the most common symptom and the most disabling symptom of Multiple Sclerosis, and its inefficient management can be a source of multiple consultations (increase in health costs) and a reduction in productivity (work stoppages).

Hence the need to define the most effective therapeutic strategy to reduce fatigue in Multiple Sclerosis.

One of the aims of this project is to provide clinical indicators that can serve as evaluation criteria for determining the most effective fatigue management strategy in Multiple Sclerosis.

The primary objective of the study is to determine the Minimal Clinically Important Difference (MCID) and the Patient Acceptable Symptomatic State (PASS) for fatigue in Multiple Sclerosis.

The source population consists of all people with Multiple Sclerosis living in Lorraine and registered in the Lorraine Registry of Multiple Sclerosis (RelSEP).

DETAILED DESCRIPTION:
Two-year patient follow-up is planned with data collection at 0, 12 and 24 months.

In addition to data already collected as part of the establishment and monitoring of the ReLSEP registry, more specific data for this study will be collected at 0, 12 and 24 months by self-questionnaires sent to patients' homes.

ELIGIBILITY:
Inclusion Criteria:

* Patient > or = 18 years old
* Patient with Multiple Sclerosis according to Mc Donald's diagnostic criteria
* Patient registered in the RelSEP registry
* Being able to fill out a questionnaire
* Person who has received complete information on the organization of the research and who has not objected to the exploitation of his data

Exclusion Criteria:

* Patients no longer residing in Lorraine
* Bedridden patients
* Patients under guardianship, curatorship or safeguard of justice
* Patients with other serious pathologies with heavy treatments (eg cancer under chemotherapy or radiotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population consists of all people with Multiple Sclerosis living in Lorraine and registered in the Lorraine Registry of Multiple Sclerosis (RelSEP).
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue score: EMIF-SEP scale | changes between 0,1 and 2 years
  measured by EMIF-SEP scale (French version of the fatigue impact scale in multiple sclerosis): 40 items and 4 dimensions (physical, psychological, cognitive, social)

SECONDARY OUTCOMES:
The quality of life: SF-36 | changes between 0,1 and 2 years
  measured by SF-36 (36-Item Short Form Survey)
The quality of life: MuSIQoL | changes between 0,1 and 2 years
  measured by MuSIQoL (Multiple Sclerosis International Quality of Life Questionnaire)
Nutritional behaviors (physical activity and sedentary lifestyle) | changes between 0,1 and 2 years
  measured by GPAQ (Global Physical Activity Questionnaire)
Psychological state (optimism, anxiety, depression) | changes between 0,1 and 2 years
  measured by HAD (Hospital Anxiety and Depression scale)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan EPSTEIN, Principal Investigator — CIC 1433 Epidémiologie Clinique Inserm, CHRU de Nancy, Université de Lorraine
Locations (1):
- CIC 1433 Épidémiologie clinique, Inserm, CHRU de Nancy, Université de Lorraine, Vandœuvre-lès-Nancy, France